CLINICAL TRIAL: NCT07079943
Title: From Adolescence to Adulthood : Analysis of the Impact of the CAPADJA Transition Support Program in Rheumatology at Bordeaux University Hospital
Brief Title: TRAJ : Transition in Rheumatology, From Adolescence to Adulthood
Acronym: TRAJ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2025/007
Record Dates: First submitted 2025-06-23; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Transitional Care
Keywords: Transitional care; Lost to follow up; Patient-reported experience; Quality of life; Patient satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAPAdJA group and Non-CAPADJA group (Other): Patients who benefited from pediatric-to-adult rheumatology transition consultation at Bordeaux University Hospital between 2017 and 2024 (Patients included 6 months after the pediatric-to-adult rheumatology transition consultation realized in the context of programm CAPADJA or not)
  Interventions: Other: Self-questionnaire : satisfaction and quality of life; Other: Self-reported questionnaire : educational or professional

INTERVENTIONS:
Other: Self-questionnaire : satisfaction and quality of life — Patient satisfaction and quality of life outcomes assessed through standardized self-reported questionnaires completed day of inclusion (6 months after the pediatric-to-adult rheumatology transition consultation realized in the context of programm CAPADJA or not. )
Other: Self-reported questionnaire : educational or professional — Patient educational or professional outcomes, assessed through standardized self-reported questionnaires completed day of inclusion (6 months after the pediatric-to-adult rheumatology transition consultation realized in the context of programm CAPADJA or not. )

SUMMARY:
This study evaluates the impact of the CAPAdJA transition support program on care continuity for young patients with chronic rheumatic diseases at Bordeaux University Hospital. The primary objective is to compare the proportion of patients lost to follow-up six months after the transition consultation between those who benefited from CAPAdJA and those who did not.

DETAILED DESCRIPTION:
The transition from pediatric to adult healthcare is a critical period for young patients with chronic diseases. This period carries risks such as disruptions in continuity of care, worsening symptoms, and a deterioration in quality of life. To address these challenges, transition support programs have been developed, including the CAPAdJA program, implemented in 2017 at Bordeaux University Hospital. While such programs seem to play a key role in structuring the transition process, their impact on care continuity and patient satisfaction remains poorly documented. The primary objective of this study is to assess the impact of the CAPAdJA program on the proportion of young patients lost to follow-up. Patients included six months after the pediatric-to-adult rheumatology transition consultation realized in the context of programm CAPADJA or not. The secondary objectives are to provide an overview of the medical and demographic characteristics of the transition in rheumatology at Bordeaux University Hospital and to analyze the impact of CAPAdJA on patient satisfaction and quality of life. Demographic and medical data will be collected using Dxcare. Then, patients will be categorized into two groups: those who benefited from the CAPAdJA support program and those who did not. Investigators will then compare the proportion of patients lost to follow-up in each group, as well as their responses to self-administered questionnaires focusing on quality of life and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients who benefited from a pediatric-to-adult rheumatology transition consultation at Bordeaux University Hospital between 2017 and 2024
* Patients over 18 years old at the time of completing the self-administered questionnaire.

Exclusion Criteria:

* Patients who do not speak French
* Patients who have refused to participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Follow-up patient | six months after the transition appointment
  The primary endpoint is the proportion of patients lost to follow-up 6 months after the transition consultation, considered to be an indicator of continuity of care and, by extension, of the medical success of the transition. This criterion will be evaluated by examining the presence or absence of follow-up consultations in the adult rheumatology department, as recorded in the CHU consultation software, six months after the transition appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier RICHER, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No